CLINICAL TRIAL: NCT05078684
Title: Ganglion Stellate Block for Treatment of Electric Storm - a Randomized Study
Brief Title: GANGlion Stellate Block for Treatment of Electric storRm (GANGSTER Trial)
Acronym: GANGSTER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Marek Sramko, MD, PhD, Head of the Department of Acute Cardiology, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-21-25
Record Dates: First submitted 2021-08-21; First posted 2021-10-14 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Ventricular Arrythmia; Ventricular Tachycardia; Ventricular Fibrillation; Arrhythmic Storm; Block
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Randomization 1:1 for active treatment vs. sham procedure
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients, attending staff, and outcome assessors will not know whether the patient received the actual LGSB or a sham (placebo) procedure. The sham procedure will consist of subcutaneous application of a small amount (1ml) of the local anesthetic drug to the region of expected LGSB procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actual LGSB (Active Comparator): The patients will receive an actual LGSB procedure:
  Using ultrasound navigation and an echo-contrast needle, 8ml of bupivacain (5%) will be applied to the site of the left ganglion stellate through an anterolateral approach in the neck region.
  Interventions: Procedure: Left ganglion stellate block
- Sham procedure (Sham Comparator): The procedure will be performed using the same instruments and anesthetic drug as the actual LGSB. However, the operator will apply only 0.5-1ml of the anesthetic drug and only subcutaneously to the site where an actual LGSB would be performed.
  Interventions: Procedure: Sham left ganglion stellate block

INTERVENTIONS:
Procedure: Left ganglion stellate block — Ultrasound-guided anesthetic block of left ganglion stellate using 8ml of 5% bupivacaine.
  Arms: Actual LGSB
Procedure: Sham left ganglion stellate block — Subcutaneous application of 0.5-1ml of 5% bupivacaine to the site of expected LGSB
  Arms: Sham procedure

SUMMARY:
This study will evaluate the acute effect of ultrasound-navigated left ganglion stellate block to suppress ventricular arrhythmia in patients with arrhythmic storm.

DETAILED DESCRIPTION:
* The study will include patients with drug-refractory arrhythmic storm indicated for left ganglion stellate block (LGSB) before or after catheter ablation.
* Included participants will be dived based on the need for mechanical ventilation and catheter ablation performed <5 days before the study
* Subsequently, the participants will be randomized to LGSB or to a sham (placebo) procedure.
* The primary endpoint will be a reduction of the burden of clinical arrhythmia >50% 24 hours after LGSB without escalation of antiarrhythmic therapy.
* The study will include 80 patients over 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. arrhythmic storm <24 hours before inclusion:

   * 3 or more episodes of sustained ventricular tachycardia (VT) or ventricular fibrillation (VF) terminated by external or internal shock,
   * or incessant VT lasting >30 minutes,
   * or very frequent nonsustained or sustained VT leading to hemodynamic instability with the need of escalation of the therapy
2. clinical indication for LBGS based on the judgment of the physician, independent of the study

Exclusion Criteria:

1. known allergy to bupivacaine
2. prior LBGS performed <7 days before the study
3. known reversible provoking trigger of the arrhythmias
4. ventricular arrhythmias triggered by premature ectopic beats during bradycardia
5. hemodynamically tolerated idiopathic VT in patients without structural heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of episodes of sustained VT/VF | 2-24 hours after LGSB. The first 2 hours after the LGSB will not be considered in the evaluation (i.e., blanking period)
  Change by >50% of the number of episodes of sustained ventricular tachycardia/fibrillation compared to 24 hours before LGSB, without escalation of antiarrhythmic therapy during 24 hours after LGSB (deep sedation requiring mechanical ventilation, addition of another antiarrhythmic drug, implantation of mechanical circulatory support, unplanned emergent catheter ablation)
Change in arrhythmia burden quantified by Holter ECG | 2-24 hours after LGSB. The first 2 hours after the LGSB will not be considered in the evaluation (i.e., blanking period)
  Change of the percent of QRS complexes with ventricular tachycardia by >50% on Holter ECG, as compared to 24 hours before LGSB, without escalation of antiarrhythmic therapy during 24 hours after LGSB (deep sedation requiring mechanical ventilation, addition of another antiarrhythmic drug, implantation of mechanical circulatory support, unplanned emergent catheter ablation).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine (IKEM), Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided